CLINICAL TRIAL: NCT02450838
Title: A Phase I Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of a Tetravalent Recombinant Subunit Dengue Vaccine (V180) in Healthy Adults Who Previously Received a Live-Attenuated Tetravalent Vaccine (TV003 or TV005)
Brief Title: Evaluating the Safety, Tolerability, and Immunogenicity of a Tetravalent Dengue Vaccine (V180) in Healthy Adults Who Previously Received a Live-Attenuated Tetravalent Vaccine (TV003 or TV005)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 301
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Dengue
Keywords: Dengue Vaccine
MeSH Terms: conditions — Dengue | interventions — Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Adjuvanted V180 vaccine (Experimental): Participants will receive one intramuscular (IM) injection of adjuvanted (with Alhydrogel™) V180 at study entry.
  Interventions: Biological: V180; Biological: Alhydrogel™
- Nonadjuvanted V180 vaccine (Experimental): Participants will receive one IM injection of nonadjuvanted V180 at study entry.
  Interventions: Biological: V180
- Placebo (Placebo Comparator): Participants will receive one IM injection of placebo at study entry.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: V180 — Tetravalent recombinant subunit dengue vaccine; V180 will contain 10 µg, 10 µg, 10 µg, and 20 µg of the DENV1, DENV2, DENV3, and DENV4 antigens, respectively.
  Arms: Adjuvanted V180 vaccine; Nonadjuvanted V180 vaccine
Biological: Alhydrogel™ — Aluminum hydroxide gel adjuvant
  Arms: Adjuvanted V180 vaccine
Biological: Placebo
  Arms: Placebo

SUMMARY:
Dengue viruses are mosquito-borne flaviviruses. Each year, dengue viruses infect millions of people throughout the tropics and subtropics. This study will evaluate the safety, tolerability, and immunogenicity of a tetravalent recombinant subunit dengue vaccine (V180) in healthy adults who previously received a live-attenuated tetravalent dengue vaccine (TV003 or TV005).

DETAILED DESCRIPTION:
Dengue fever is caused by any one of four viral serotypes (DENV1, DENV2, DENV3, and DENV4) and infection by any serotype creates life-long immunity against that serotype. V180 is an experimental tetravalent recombinant subunit dengue vaccine that would protect against all four serotypes (DENV1, DENV2, DENV3, and DENV4). The purpose of this study is to evaluate the safety, tolerability, and immunogenicity of adjuvanted (with Alhydrogel™) and nonadjuvanted formulations of V180 in healthy adults who have previously received the live-attenuated tetravalent dengue vaccine TV003 or TV005.

Participants will be randomly assigned to receive one intramuscular injection of either adjuvanted V180, nonadjuvanted V180, or placebo at study entry (Day 1). Participants will record their temperature and any adverse events for 14 days after receiving the vaccination. Additional study visits will occur on Days 15, 28 and 180. Visits will include a physical examination and blood and urine collection. Study staff will contact participants by telephone at Days 7 and 90 (and at other occasional time points between Days 90 and 180) for health and safety follow-up monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female between 18 and 50 years of age, inclusive
* Has previously received TV003 or TV005 live-attenuated tetravalent vaccine (LATV) DENV vaccine, successfully completed the study with no safety concerns, and seroconverted to 3 or more serotypes
* Good general health as determined by physical examination, laboratory screening, and review of medical history
* Willingness to participate in the study as evidenced by signing the informed consent document
* Willingness to complete all scheduled visits and to comply with the study procedures
* Available for the duration of the study, approximately 26 weeks post-vaccination
* Ability to read, understand, and complete study questionnaires (i.e., the Vaccination Report Card)
* Has access to a telephone
* Is afebrile (less than 100.4°F [less than 38.0°C] oral or equivalent) for 72 hours prior to vaccination. Note: If a participant is not afebrile for 72 hours prior to vaccination, vaccination can be deferred if all other eligibility criteria are met and time allows for vaccination.
* Females Only: Female participants of childbearing potential willing to use effective contraception for the duration of the trial. Reliable methods of contraception include: hormonal birth control, condoms with spermicide, diaphragm with spermicide, surgical sterilization, intrauterine device, and abstinence (6 months or longer since last sexual encounter). All female participants will be considered having childbearing potential except for those with hysterectomy, tubal ligation, tubal coil (at least 3 months prior to vaccination), or post-menopausal status documented as at least 1 year since last menstrual period.

Exclusion Criteria:

* Is pregnant or breastfeeding, or expecting to conceive at any time from signing the informed consent through Day 180 after receiving the study vaccine/placebo
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the requirements of the study protocol
* Has 1 or more of the following screening laboratory values:

  1. Alanine aminotransferase (ALT) greater than or equal to 1.25 times the upper limit of normal (ULN)
  2. Positive urine glucose or urine protein greater than 1+ by dipstick or urinalysis
  3. Serum creatinine greater than ULN by gender
  4. Hematology results as follows:

     * Hemoglobin meeting Grade 1 or higher criteria
     * Absolute neutrophil count (ANC) less than 1,000/mm^3
     * Platelets less than or equal to 140,000/mm^3
* Any significant alcohol or drug abuse within 12 months prior to screening which has caused medical, occupational, or family problems, as indicated by participant history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the last 6 months)
* Any known immunodeficiency syndrome. (Participant has known, suspected, or a history of immunocompromise, including congenital immunodeficiency, human immunodeficiency virus (HIV) infection, leukemia, lymphoma, Hodgkin's disease, multiple myeloma, generalized malignancy, chronic renal failure (most recent serum creatinine values in medical record greater than or equal to 3 mg/dL), nephrotic syndrome, or other conditions associated with immunosuppression, including ever receiving organ or bone marrow transplant.)
* Hepatitis C virus (HCV) infection, by screening and confirmatory assays
* Hepatitis B virus (HBV) infection, by hepatitis B surface antigen (HBsAg) screening
* Use of anticoagulant medications
* Known or suspected impairment of immunological function
* Has received systemic corticosteroids (equivalent of greater than or equal to 2 mg/kg total daily dose of prednisone or greater than or equal to 20 mg/d for persons weighing greater than 10 kg) for greater than or equal to 14 consecutive days and has not completed treatment at least 30 days prior to study entry, or plans to receive these systemic corticosteroids 28 days following vaccination
* Has received systemic corticosteroids exceeding physiologic replacement doses (~5 mg/d prednisone equivalent) within 14 days prior to vaccination, or plans to receive these systemic corticosteroids 28 days following vaccination
* Has received immunosuppressive therapies including chemotherapeutic agents used to treat cancer or other conditions, and treatments associated with organ or bone marrow transplantation, or autoimmune disease, or plans to receive these immunosuppressive therapies 28 days following vaccination
* Has received a licensed non-live vaccine within 14 days prior to receipt of the first dose of study vaccine/placebo, or plans to receive a licensed non-live vaccine at any time from receiving the first dose of study vaccine/placebo through 28 days after receiving the last dose of the study vaccine/placebo (Exception: Inactivated influenza vaccine may be administered during the study, but must be given at least 7 days prior to receipt of the study vaccine/placebo or at least 15 days after receipt of the study vaccine/placebo.)
* Has received a licensed live vaccine within 30 days prior to receipt of the first dose of study vaccine/placebo, or plans to receive a licensed live vaccine at any time from receiving the first dose of study vaccine/placebo through 28 days after receiving the last dose of the study vaccine/placebo.
* Asplenia
* Receipt of blood products within the past 6 months prior to receipt of study vaccine or placebo, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin at any time from signing the informed consent through 28 days post-vaccination
* History of flavivirus infection or vaccination in the interim since receipt of the last dose of the experimental dengue vaccine (TV003 or TV005) (e.g., wild type dengue, yellow fever virus, St. Louis encephalitis virus, West Nile virus (WNV), Japanese encephalitis virus, tick-borne encephalitis virus)
* History of travel to a flavivirus endemic area in the interim since receipt of the last dose of the experimental dengue vaccine (TV003 or TV005), with evidence of a flavivirus exposure as documented by appropriate screening in accordance with the country of travel
* Serological evidence of WNV infection since receipt of last dose of experimental dengue vaccine (TV003 or TV005), as evidenced by a greater than or equal to 4-fold rise in titer using paired serum. Serum from the last study visit since receipt of TV003 or TV005 will be paired from serum collected at screening.
* Anticipated receipt of any investigational agent in the 42 days prior to signing the informed consent, or plans to receive such products (other than the study vaccine/placebo) at any time during enrollment in this clinical study
* Has definite plans to travel to a dengue endemic area in the 30 days before or anytime during the study
* Refusal to allow storage of specimens for future research
* History of febrile illness (greater than or equal to 100.4°F [greater than or equal to 38.0°C] oral or equivalent) occurring within 72 hours prior to receipt of the first dose of study vaccine/placebo. Note: If a participant is febrile within 72 hours prior to vaccination, vaccination can be deferred if all other eligibility criteria are met and time allows for vaccination.
* Known hypersensitivity to any component of the dengue vaccine, known hypersensitivity to an aminoglycoside antibiotic, or history of severe allergic reaction (e.g., swelling of the mouth and throat, difficulty breathing, hypotension or shock) that required medical intervention
* Has a history of malignancy less than or equal to 5 years prior to signing informed consent
* Has poorly controlled diabetes mellitus, is receiving insulin or an oral antidiabetic agent, and has a glycosylated hemoglobin (HbA1c) level greater than or equal to 9% (greater than or equal to 3.5% ULN) tested within 28 days of vaccination. Note: For those participants who report a medical history of diabetes mellitus during screening, and cannot provide an HbA1c level within 28 days prior to screening, perform HbA1c level to assess whether participant is excluded from the study based upon this criterion.
* Planned donation of eggs or sperm at any time from signing the informed consent through 28 days after receiving the last dose of the study vaccine/placebo
* Recent hospitalization for acute medical illness within the 3 months prior to receipt of study vaccine/placebo (exception: minor trauma)
* Has previously failed screening for this study and was not eligible for rescreening
* Has previously been enrolled into this study and subsequently withdrawn
* Is unlikely to adhere to study procedures, keep appointments, or is planning to relocate during the study
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is investigational site or SPONSOR staff directly involved with this trial
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Virus neutralizing antibody levels, as measured by the PRNT with a 50% neutralization cutoff (PRNT50 titer) | Measured at Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research (CIR), Johns Hopkins School of Public Health; Kristen Pierce, MD, Principal Investigator — University of Vermont
Locations (3):
- United States (3):
  - Center for Immunization Research, Johns Hopkins School of Public Health, Baltimore, Maryland
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont Vaccine Testing Center, Burlington, Vermont